CLINICAL TRIAL: NCT04661982
Title: Long Term Follow Up After Breast Cancer
Brief Title: Long Term Follow-Up in Patients With Stage 0-IIIC Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07100; NCI-2019-03481 (Other: Registry ID: CTRP (Clinical Trial Reporting Program)); 07100 (Other: City of Hope Medical Center)
Record Dates: First submitted 2012-02-09; First posted 2020-12-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor, lymph node, blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (long term follow-up): Patients undergo long term follow-up and complete questionnaires.
  Interventions: Other: Long-term Follow-up; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Long-term Follow-up — Undergo long term follow-up
  Other Names: LONG-TERM FOLLOW-UP, Long-term Follow-up
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This trial studies long term follow-up care in patients with stage 0-IIIC breast cancer. Collecting feedback from breast cancer patients may help researchers to define comprehensive long term follow-up care for breast cancer survivors, better understand health-related quality of life and long-term complications in breast cancer survivors, and to increase the knowledge of the mechanisms by which a patient's own immune system attempts to combat breast cancer, and what factors may make this response more successful.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide comprehensive care to breast cancer survivors diagnosed with stage 0 to IIIC, who received at least part of their treatment at City of Hope.

II. To use the information obtained from follow-up of breast cancer survivors to describe the magnitude of risk and associated risk factors.

III. To use the information gained from follow-up of breast cancer survivors to describe health-related quality of life (HRQL) concerns in breast cancer survivors and identify those at highest risk.

OUTLINE:

Patients undergo long term follow-up and complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer, stage 0-IIIC
* Partial or entire treatment at City of Hope
* Must be registered before adjuvant therapy and ideally before definitive local therapy

Exclusion Criteria:

* Stage IV breast cancer
* Recurrent breast cancer
* Prior cancers, chemotherapy or radiation * (Note: Subjects who develop locoregional or systemic recurrence while enrolled on this protocol will be withdrawn, and will continue their care with their primary oncology providers only)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stage 0-IIIC breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-07-06 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
Incidence rates of the study end-points | Up to 12 years
  Will estimation of incidence rates of the study end-points that may be associated with original diagnosis or treatment received, and delineation of temporal changes in serial measurements and their relationship to time-invariant characteristics such as original diagnosis, race, and education and time varying characteristics such as age and body mass index (BMI). Incidence rates may be compared with national standards adjusted for key demographic variables and between patient subgroups. Time of entry onto the study in the analysis will be from the date of diagnosis of primary disease. Stepwise logistic regression analysis of endpoints of interest at certain follow-up time may be conducted, accounting for the joint effect of such factors as age, time since diagnosis and treatment, radiation dose, chemotherapy and tumor subtype.
FACT- Cog | Change from pre-treatment baseline over a 2-year period
  Functional Assessment of Cancer Therapy Cognitive Function
Cancer induced immune dysfunction | Up to 12 years
  Will analyze patients' tumor, lymph node, and blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States